CLINICAL TRIAL: NCT00988819
Title: Developmental Pathways to Metabolic Diseases: Metabolic Physiology, Epigenetics and Body Composition in Healthy Overweight and Obese Subjects With a Fixed Range of Body Mass Index in Singapore - To Investigate the Influence of Ethnicity
Brief Title: To Investigate the Influence of Ethnicity in Metabolic Disease in Healthy, Overweight and Obese Subjects
Acronym: SAMS-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Associate Professor Chong Yap Seng, National University of Singapore (NUHS)
Other Study IDs: DSRB C/09/022
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Healthy; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, packed cells, blood clot, urine, buccal cells, muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The overall objective of this study is to investigate in depth the nature of metabolic physiology, body composition and epigenetic differences of the different phenotypes of overweight and obese individuals who are otherwise overtly healthy among the three major ethnic groups in Singapore.

DETAILED DESCRIPTION:
Over the past decade, investigators in Singapore have been actively studying the impact of ethnicity on metabolic traits, particularly those related to insulin resistance (detailed in the preliminary data of this proposal. We have observed that, for the same BMI, Asian Indians appear to have greater insulin resistance than Chinese. In line with the greater insulin resistance observed in Asian Indians, it has also been noted that Asian Indians exhibit greater central obesity (manifest as a larger waist circumference). In some ways, this resembles the phenotype that might be expected if the mismatch pathway described in this proposal, were involved in the pathogenesis of insulin resistance in this ethnic group. Interestingly, Asian Indians have also been noted to have lower birth weight than Chinese in our population. In contrast, although Malays are more insulin resistant than Chinese, this is largely due to greater adiposity and, after adjustment for body mass index, Malays are actually less insulin resistant than their Chinese and Asian Indian counterparts. They also have smaller waist circumferences. It is also recognized that pregnant Malay women tend to be generally more obese than their Chinese and Asian Indian counterparts, which may put their children at great risk of fetal hyperinsulinemia. As such, the potential exists that this latter pathway is more active in the pathogenesis of insulin resistance in this ethnic group.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Chinese, Malay or Indian males (aged 21-40)
3. Body mass index between 23-30 kg/m2 for the overweight or obese subjects and between 18.5 to 22.9 kg/m2 for the Chinese control group
4. Sedentary adults < 1 episode of exercise > =30 min/week
5. Birth weight between 3-97% percentiles
6. Fasting glucose < 7 mmol/L
7. Normotensive, defined as BP < 140/90 mmHg and not on any antihypertensive agents

Exclusion Criteria:

1. Recent changes in weight of > 5% over the past 6 months
2. Attempts to lose weight (weight not reaching equilibrium, exercises still changing and not in maintenance phase) over the past 6 months
3. Significant changes in diet over the past 6 months
4. Any use of weight reducing drugs in the past 6 months
5. Previous abdominal surgery (and bariatric surgery)
6. Any bleeding disorders which would preclude biopsies
7. Any use of investigational drugs in the past 6 months
8. Known allergy to insulin or local anesthetics
9. Known allergy to milk or milk products (eg. Ensure)
10. Any serious illness requiring hospitalization or surgery in the past 6 months
11. Treatment with medications for hypertension, diabetes mellitus or dyslipidemia, epilepsy, ischemic heart disease
12. On anti-platelet agents, non-steroidal anti-inflammatory drugs (NSAIDs) or anticoagulants
13. Use of any prescription medication that cannot be safely discontinued within 14 days prior to study entry
14. Any use of corticosteroids in the past 6 months
15. Any other medications that could alter insulin resistance
16. History of surgery with metallic clips, staples or stents
17. Presence of cardiac pacemaker or other foreign body in any part of the body
18. Mother no longer alive or unable to provide information on birth weight
19. Born premature (ie. not full term baby < 37 weeks of gestation age)

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Singapore population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Overall Officials: E Shyong Tai, Principal Investigator — National University Hospital, Singapore; Yung Seng Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan ALM, Langley SR, Tan CF, Chai JF, Khoo CM, Leow MK, Khoo EYH, Moreno-Moral A, Pravenec M, Rotival M, Sadananthan SA, Velan SS, Venkataraman K, Chong YS, Lee YS, Sim X, Stunkel W, Liu MH, Tai ES, Petretto E. Ethnicity-Specific Skeletal Muscle Transcriptional Signatures and Their Relevance to Insulin Resistance in Singapore. J Clin Endocrinol Metab. 2019 Feb 1;104(2):465-486. doi: 10.1210/jc.2018-00309. PMID 30137523
- [Derived] Lee Y, Chong MF, Liu JC, Libedinsky C, Gooley JJ, Chen S, Wu T, Tan V, Zhou M, Meaney MJ, Lee YS, Chee MW. Dietary disinhibition modulates neural valuation of food in the fed and fasted states. Am J Clin Nutr. 2013 May;97(5):919-25. doi: 10.3945/ajcn.112.053801. Epub 2013 Apr 3. PMID 23553164